CLINICAL TRIAL: NCT00822692
Title: Prospective Randomized Double Blind, Placebo-Controlled Trial of Septra for Uncomplicated Skin Abscesses in Patients at Risk for Community Acquired Methicillin-Resistant Staphylococcus Aureus Infection on 30 Day Recurrence Rates.
Brief Title: Trial of Septra for Uncomplicated Skin Abscesses in Patients at Risk for Community Acquired Methicillin-Resistant Staphylococcus Aureus Infection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 59th Medical Wing (U.S. Federal Agency)
Collaborators: U.S. Air Force Office of the Surgeon General (U.S. Federal Agency); Emergency Medicine Foundation (Other)
Responsible Party: Principal Investigator, Gillian Schmitz, Emergency Physician, 59th Medical Wing
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FWH20080055H
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2009-09-03 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-12

CONDITIONS: Abscess; Methicillin-Resistant Staphylococcus Aureus Infection
Keywords: Abscess; Cellulitis; Antibiotics; MRSA
MeSH Terms: conditions — Abscess; Cellulitis | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bactrim DS (Active Comparator): Trim/sulfa (800/160) two tablets orally (PO) twice a day (BID) x 7 days
  Interventions: Drug: Trim/ Sulfa DS
- matched placebo (Placebo Comparator): matched placebo 2 pills orally (PO) twice a day (BID) x 7 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Trim/ Sulfa DS — bactrim DS (800/160) two tablets PO BID x 7 days
  Other Names: Bactrim
  Arms: Bactrim DS
Drug: placebo — matched placebo 2 pills PO BID x 7 days
  Arms: matched placebo

SUMMARY:
Patients will be enrolled in a multi-center study (Wilford Hall Medical Center and Brooke Army Medical Center) to prospectively evaluate outcome after treatment for an uncomplicated skin abscess.

DETAILED DESCRIPTION:
All patients will receive incision and drainage and wound cultures. Patients will then be randomized to 1) septa double strength two pills orally twice a day x 7 days or 2)placebo. Patients will then return to the emergency room on days 3 and 7 for wound repacking and evaluation. The primary outcome recurrence rates within 30 days of treatment. Patients who are not improving at the following visit will then be treated with additional antibiotics if needed. Data will be analyzed both by initial randomization and intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18-65 who present to the emergency department with a skin abscess that requires incision and drainage.

Exclusion Criteria:

* Patients with diabetes, HIV, cancer or other immunocompromised patients.
* Additionally, any patients who received antibiotics within one week of presentation or were hospitalized in previous month will be excluded to minimize potential confounding variables.
* Pregnant and breastfeeding patients will also be excluded due to possible safety concerns with antibiotic treatment.
* Patients with abscesses on head, face, perirectal, or periananal regions, abscesses with known tracks or fistulas to deeper structures, or abscesses requiring surgical drainage in an operating room are excluded.
* Finally, patients with sulfa allergy will be excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2008-07; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gillian R Schmitz, Principal Investigator — 59th Medical Wing
Locations (1):
- Wilford Hall Medical Center, Lackland Air Force Base, Texas, United States

REFERENCES:
- [Derived] Schmitz GR, Bruner D, Pitotti R, Olderog C, Livengood T, Williams J, Huebner K, Lightfoot J, Ritz B, Bates C, Schmitz M, Mete M, Deye G. Randomized controlled trial of trimethoprim-sulfamethoxazole for uncomplicated skin abscesses in patients at risk for community-associated methicillin-resistant Staphylococcus aureus infection. Ann Emerg Med. 2010 Sep;56(3):283-7. doi: 10.1016/j.annemergmed.2010.03.002. Epub 2010 Mar 26. PMID 20346539

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at 3 hospital emergency departments from July 1, 2008 to June 1, 2009.
Pre-assignment Details: Patients were assigned by block randomization and data was analyzed with intention to treat analysis.
Groups:
- Bactrim DS (800/160) Two Tablets PO BID x 7 Days: Active Intervention Arm
- Matched Placebo 2 Pills PO BID x 7 Days: Placebo arm
Period: Overall Study
Arm/Group | Bactrim DS (800/160) Two Tablets PO BID x 7 Days | Matched Placebo 2 Pills PO BID x 7 Days
Started | 63 (July 1, 2008) | 76 (July 1, 2008)
Completed | 46 (June 1, 2009) | 51 (June 1 , 2009)
Not Completed | 17 | 25
Not completed — Lost to Follow-up | 17 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bactrim DS (800/160) Two Tablets PO BID x 7 Days | Matched Placebo 2 Pills PO BID x 7 Days | Total
Number analyzed (Participants) | 63 | 76 | 139
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 63 | 76 | 139
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (13) | 30.6 (13) | 31.06 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 35 | 53
  Male | 45 | 41 | 86
Region of Enrollment [Number; unit: participants]
  United States | 63 | 76 | 139

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Rates of Abscesses
Description: Number of patient with a new abscess in same or different location as previous lesion
Time Frame: 30 days after incision and drainage
Measure: Number; unit: participants
Arm/Group | Bactrim DS (800/160) Two Tablets PO BID x 7 Days | Matched Placebo 2 Pills PO BID x 7 Days
Number analyzed (Participants) | 46 | 51
participants | 4 | 14

ADVERSE EVENTS:
Groups:
- Bactrim DS (800/160) Two Tablets PO BID x 7 Days: bactrim DS (800/160) two tablets PO BID x 7 days
- Matched Placebo 2 Pills PO BID x 7 Days: matched placebo 2 pills PO BID x 7 days
Arm/Group | Bactrim DS (800/160) Two Tablets PO BID x 7 Days | Matched Placebo 2 Pills PO BID x 7 Days
Serious Adverse Events (participants affected / at risk) | 0/63 | 0/76
Other Adverse Events (participants affected / at risk) | 15/63 | 27/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bactrim DS (800/160) Two Tablets PO BID x 7 Days (N=63) | Matched Placebo 2 Pills PO BID x 7 Days (N=76)
treatment failure (Skin and subcutaneous tissue disorders) | 15 | 27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No